CLINICAL TRIAL: NCT02145793
Title: Exploring the Group Visit Model for Pediatric ADHD Management in the Medical Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Nerissa Bauer, Assistant Professor, Indiana University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1204008526
Record Dates: First submitted 2014-05-18; First posted 2014-05-23 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: ADHD
Keywords: primary care; pediatrics; parenting; education
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ADHD Group Curriculum (Active Comparator): Participants assigned to the group visit intervention agree to participate in 5 group visits every 3 months rather than individual ADHD follow-up visits to the clinic. Parents and children participate in separate but simultaneously run groups. Group portion is 60 minutes and then parent-child dyads complete individual visits for medication titration and physical exam.
  Interventions: Behavioral: ADHD Group Curriculum
- Control (No Intervention): Participants continue to go to the clinic for 5 routine ADHD follow-up visits to the clinic every 3 months as usual clinical protocol.

INTERVENTIONS:
Behavioral: ADHD Group Curriculum — Study specific ADHD Group curriculum was designed and implemented for the study. Parent curriculum included the following topics: What is ADHD, medications, educational advocacy, how to prevent behavioral issues and how to defuse common behavioral challenges and manage stress. Child curriculum included the following topics: what is ADHD, social skills and friendships, handling school and organization skills, understanding feelings and managing negative emotions
  Arms: ADHD Group Curriculum

SUMMARY:
Attention deficit hyperactivity disorder (ADHD) affects 8% of US youth. Even though evidence shows medications are effective in reducing ADHD symptoms, many families experience ongoing parenting stress around parent-child interactions. Children often have ongoing impairments in functioning. ADHD is a common condition identified and managed by primary care pediatricians. However current care in the clinic is not optimal to address parents' and children's needs around ADHD chronic care. Time is the biggest barrier. Group visits are a viable option to improve pediatric ADHD care, but requires extensive study. The goal of this proposed study is to test the feasibility and effectiveness of the group visit model for ADHD management within pediatric primary care. This study will be a randomized feasibility study that will generate important pilot data, as well as result in an innovative, exportable pediatric ADHD group curriculum for primary care practice.

DETAILED DESCRIPTION:
The specific research aims of this proposal are:

Aim 1: Develop and test a group curriculum for parents of children (age 6 to 18 years) with ADHD to increase parental knowledge about ADHD and self-confidence in managing issues related to their child's functioning in school and home.

Aim 2: Develop and test a group curriculum for children (age 6 to 18 years) with ADHD to teach social and educational skills to improve adaptive functioning at home and school.

Aim 3: To assess any added benefits to the parents, children and providers (related to group visit logistics and satisfaction) the group visit model has over usual care.

Aim 4: To assess whether the group visit model can be done efficiently and effectively in the setting of an actual general pediatric practice.

ELIGIBILITY:
Inclusion Criteria:

* children with ADHD and their parents
* children receiving routine ADHD follow-up care at the study clinic
* if on medication, must be "stable" for 3 months and therefore not needing monthly clinic appointments to titrate medication

Exclusion Criteria:

* conduct disorder
* autism
* moderate to severe intellectual disability

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2012-06; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Number of clinic visits during study period | 12 months
  Feasibility of group visit model was measured as number of visits to the clinic by chart review. We also looked at the number of group visits a family attended based on the sign in sheet provided at the beginning of each session.

SECONDARY OUTCOMES:
Parent-rated ADHD symptoms | Baseline
  Parents completed validated Vanderbilt Rating Scale regarding child's ADHD symptoms. Measures response to ADHD treatment, primarily medication.
Parent-rated ADHD symptoms | 12 months
  Parents complete validated Vanderbilt Rating Scale to report child symptoms of ADHD. Used to assess response to treatment, usually medication.
Child functioning at home | Baseline
  Parent report of adaptive functioning of child in the home setting using the Home Situations Questionnaire
Child functioning at home | 12 months
  Parents report of child's adaptive functioning in the home setting using the Home Situations Questionnaire.
Teacher report of child's ADHD symptoms | baseline
  teachers received the validated Vanderbilt rating scale to rate student's ADHD symptoms in the classroom. Parents were given the tool at time of enrollment and asked to give to teacher as per clinical care guidelines. Monitors impact of ADHD treatment, usually medication.
teacher report of child's ADHD symptoms in school | 12 months
  teachers received the validated Vanderbilt rating scale to rate student's ADHD symptoms in the classroom. Parents were given the tool at time of enrollment and asked to give to teacher as per clinical care guidelines. Monitors impact of ADHD treatment, usually medication.
Child functioning at school | baseline
  teachers were invited to provide rating of child's adaptive functioning at school. Parent given the tool at time of enrollment and instructed to give to teacher as per clinical care guidelines.
teacher rating of child's functioning in school | 12 months
  teachers were invited to provide rating of child's adaptive functioning at school. Parent given the tool at time of enrollment and instructed to give to teacher as per clinical care guidelines.
Quality of Life | baseline
  Capture parent rating of quality of life related to ADHD using the Child Health Questionnaire-28 validated tool.
Quality of Life | 12 months
  Capture parent rating of quality of life related to ADHD using the Child Health Questionnaire-28 validated tool.
Parenting self-efficacy | Baseline
  Parent reported sense of confidence using the Parenting Sense of Confidence Scale
Parenting Self-efficacy | 12 months
  Parent-reported sense of confidence using Parenting Sense of Confidence scale
Parental knowledge, satisfaction towards medication treatment | baseline
  Parent report of knowledge, attitudes and satisfaction towards medication experiences with ADHD medication treatment
Parent knowledge and satisfaction towards medication treatment | 12 months
  Parent report of knowledge, attitudes and satisfaction towards medication experiences with ADHD medication treatment

OTHER OUTCOMES:
Participant feedback about the curriculum | after each group visit over 365 days
  parents and children separately complete a short 4 question survey about what they liked, what they did not like, what they are excited about doing after the group visit and suggestions for improvement. Data used to continually refine the curriculum. At the 5th group visit, participants participated in informal discussion about the group visit model and overall satisfaction with the intervention
Pediatric facilitator and staff feedback | at the end of each group visit over 365 days
  collected informal feedback and reflection about the process, barriers and positive experiences overall about the group visit model and impact on the clinical workflow, suggestions for improvement that was used to continually refine the model for quality improvement

CONTACTS AND LOCATIONS:
Overall Officials: Nerissa S Bauer, MD, MPH, Principal Investigator — Indiana University School of Medicine
Locations (1):
- General Pediatrics Clinic Medical Service Area 1 in Riley Hospital for Children at IU Health, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Bauer NS, Szczepaniak D, Sullivan PD, Mooneyham G, Pottenger A, Johnson CS, Downs SM. Group Visits to Improve Pediatric Attention-Deficit Hyperactivity Disorder Chronic Care Management. J Dev Behav Pediatr. 2015 Oct;36(8):553-61. doi: 10.1097/DBP.0000000000000207. PMID 26414089